CLINICAL TRIAL: NCT03182530
Title: Prevention of Radial Artery Occlusion After Trans-radial Cardiac Catheterization. Randomized Duplex Follow-up Study.
Brief Title: Prevention of Radial Artery Occlusion After Trans-radial Cardiac Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Abbas Abdelaal, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRCC
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: CARDIAC CATHETRIZATION

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ULTRA method group (Active Comparator)
  Interventions: Device: ulnar artery compression device; Device: radial artery compression device
- standard patent hemostasis group (Active Comparator)
  Interventions: Device: radial artery compression device guided with plysthmography
- control group (Experimental)
  Interventions: Device: radial artery compression device

INTERVENTIONS:
Device: ulnar artery compression device — a radial compression device will be applied at the access site. another closure device will be used for ipsilateral ulnar artery compression for 1-hour duration in order to increase peak velocity blood flow into the radi¬al artery. neither pulse oxymetry nor duplex ultrasonography will be performed in case of ulnar artery compression. after ulnar artery compression, the initial compression of the radial artery will be reduced by letting up the pressure until bleeding will be seen and then adding minimal pressure whenever needed in order to maintain radial artery patency.
  Arms: ULTRA method group
Device: radial artery compression device guided with plysthmography — a radial compression device will be applied at the access site. A pulse oximeter sensor was placed over the index finger. Transient ipsilateral ulnar artery will be occluded manually to evaluate the status of radial artery patency by plethysmography (digital pulse analysis), and if there's lack of signal, the process of deflation and reinflation of the radial artery device's bladder will be repeated over the next 15 min to attempt re-establishment of antegrade radial artery flow without affecting hemostasis
  Arms: standard patent hemostasis group
Device: radial artery compression device — patients undergo the conventional hemostasis compression by using a radial compression device applied at the access site.
  Arms: ULTRA method group; control group

SUMMARY:
Data from literature: transradial access failure sometimes occurs due to inability to cannulate the radial artery due to radial artery spasm1 causing severe difficulties in manipulation of the guide wires and catheters along the tortuous pathways of the arteries. both mechanical stimuli and circulating catecholamines through activation of α1-adrenoreceptors, causing smooth muscle cell contraction & radial artery spasm

ELIGIBILITY:
Inclusion Criteria:

* Normal radial artery and of size ≥ 2mm by duplex.
* Normal ulnar artery by duplex.

Exclusion Criteria:

* Pre-procedural duplex detection of radial artery anomalies as hypoplasia, tortousity, severe calcification or radial artery diameter < 2 mm.
* Severe renal failure (creatinine clearance < 30 ml/min).
* Known peripheral vascular disease.
* Emergency procedures.
* Failure to successfully cannulate the radial artery was also a criterion for exclusion.
* Patients on warfarin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The percentage of occurrence of radial artery occlusion | 1 hour
  the assessment will be done after compression device removal guided by duplex post trans-radial cardiac catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek nagib, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No